CLINICAL TRIAL: NCT03973307
Title: Evaluation of UroX™ Biomarker Screening Test in the Investigation of Bladder Cancer From Urine Samples - a Single Site Pilot Study
Brief Title: UroX Biomarker Bladder Cancer Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: KDx Diagnostics Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD2018-68
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with bladder cancer: 50 participants with histologically confirmed evidence of malignancy for bladder cancer following routine cystoscopy and biopsy.
  Interventions: Diagnostic Test: UroX bladder cancer biomarker test
- Participants without bladder cancer: 50 participants with negative biopsy for bladder cancer following routine cystoscopy and biopsy.
  Interventions: Diagnostic Test: UroX bladder cancer biomarker test

INTERVENTIONS:
Diagnostic Test: UroX bladder cancer biomarker test — Urine test using novel UroX biomarker test for bladder malignancy

SUMMARY:
This is a prospective observational study looking at urine samples from participants under referral for a standard of care investigative cystoscopy and biopsy.

The study aims to test if the UroX™ biomarker (a measurable indicator of a biological condition) can be detected in urine samples from participants who may later test positive following a biopsy for bladder cancer. The study aims to assess the value of the biomarker as a screening tool for bladder cancer.

Patients with and those without bladder cancer are required for the study.

DETAILED DESCRIPTION:
Patients who undergo investigation for bladder cancer will have a cystoscopy and biopsy as part of their routine care. These patients are then brought back to urology outpatient clinic for their biopsy results within two weeks.

A UroX Biomarker Bladder Cancer Study patient information leaflet will be sent to all patients who are booked for these investigations, explaining the study aims and the requirements for participation.

On the day of their cystoscopy, potential participants will be approached and after signing a study specific consent form, the urine sample will be accepted, given a study number and sent for UroX biomarker testing.

These results will then be returned to the study team for comparison against the biopsy histology result to assess for sensitivity and specificity.

While cystoscopy and biopsy are the current gold standard for diagnosis of bladder cancer, it has been shown to have false-negatives of between 10-40%, due to factors such as operator error or small areas of malignancy(15-17). The possibility of a screening/outpatient test for bladder cancer with high positive predictive value would help with reduction or prioritisation of further investigations and early diagnosis of disease thus potentially allowing alternative treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years of age
* Patients under investigation for bladder cancer due to undergo investigative standard of care biopsy

Exclusion Criteria:

* Patients aged < 18 years of age
* Patients who are currently undergoing radiation therapy.
* Proposed subject has no bladder (due to surgical removal).
* No cystoscopy and/or pathology information for proposed subject (following cystoscopy for final inclusion in study results)
* Patients unable or unwilling to provide consent
* Patients currently on investigational drug trials
* Patients with Catheter in Situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants under investigation for possible bladder cancer due to undergo cystoscopy and biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy of the UroX™ biomarker urine test | 1 day (single visit/test)
  UroX™ urine biomarker staining result compared with standard of care biopsy result

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Vasdev, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No